CLINICAL TRIAL: NCT02046070
Title: An Open-Label, Phase 2 Study to Evaluate the Oral Combination of Ixazomib (MLN9708) With Cyclophosphamide and Dexamethasone in Patients With Newly Diagnosed or Relapsed and/or Refractory Multiple Myeloma Requiring Systemic Treatment
Brief Title: Phase 2 Study to Evaluate the Oral Combination of Ixazomib (MLN9708) With Cyclophosphamide and Dexamethasone in Patients With Newly Diagnosed or Relapsed and/or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C16020; 2013-003113-17 (EudraCT Number); U1111-1158-2714 (Registry Identifier: WHO)
Record Dates: First submitted 2013-12-12; First posted 2014-01-27 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-06

CONDITIONS: Multiple Myeloma
Keywords: MLN9708; Newly diagnosed; NDMM; IXAZOMIB; RRMM
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; ixazomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) (Experimental): Ixazomib 4.0 mg, capsules, orally, on Days 1, 8, 15 of a 28-day cycle until progressive disease (PD)/death or unacceptable toxicity [13 cycles in the Induction Phase continuing in the Maintenance Phase for up to 36 Months] and cyclophosphamide (CYC) 300 mg/m^2, tablets, orally, on Days 1, 8 and 15 of a 28-day cycle for 13 cycles or until PD/death or unacceptable toxicity and dexamethasone (DEX) 40 mg, tablets, orally, on Days 1, 8, 15 and 22 (dose reduced to 20 mg for patients >75 years) of a 28-day cycle for 13 cycles or until PD/death or unacceptable toxicity in participants with NDMM.
  Interventions: Drug: Cyclophosphamide; Drug: Ixazomib; Drug: Dexamethasone
- Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM) (Experimental): Ixazomib 4.0 mg, capsules, orally, on Days 1, 8, 15 of a 28-day cycle until PD/death or unacceptable toxicity [13 cycles in the Induction Phase continuing in the Maintenance Phase for up to 36 Months] and cyclophosphamide (CYC) 400 mg/m^2, tablets, orally, on Days 1, 8 and 15 of a 28-day cycle for 13 cycles or until PD/death or unacceptable toxicity and dexamethasone (DEX) 40 mg, tablets, orally, on Days 1, 8, 15 and 22 (dose reduced to 20 mg for patients >75 years) of a 28-day cycle for 13 cycles or until PD/death or unacceptable toxicity in participants with NDMM.
  Interventions: Drug: Cyclophosphamide; Drug: Ixazomib; Drug: Dexamethasone
- Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM) (Experimental): Ixazomib 4.0 mg, capsules, orally, on Days 1, 8, 15 of a 28-day cycle and cyclophosphamide 300 mg/m^2, tablets, orally, on Days 1, 8 and 15 of a 28-day cycle and dexamethasone (DEX) 40 mg, tablets, orally, on Days 1, 8, 15 and 22 (dose reduced to 20 mg for patients >75 years) of a 28-day cycle until PD/death or unacceptable toxicity in participants with RRMM.
  Interventions: Drug: Cyclophosphamide; Drug: Ixazomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide tablets
Drug: Ixazomib — Ixazomib capsules
  Other Names: MLN9708
Drug: Dexamethasone — Dexamethasone tablets

SUMMARY:
This is a phase 2, multicenter, open-label study in patients with Newly Diagnosed Multiple Myeloma (NDMM) who have not received prior systemic treatment for multiple myeloma (MM) and who are ineligible for high-dose therapy (HDT)-stem cell transplantation (SCT) due to age (ie, ≥ 65 years) or comorbid disease(s) or with Relapsed and/or Refractory Multiple Myeloma (RRMM).

DETAILED DESCRIPTION:
The investigational drug being tested in this study is called MLN9708 also known as Ixazomib. This study will look at disease response rates and safety in people who take ixazomib in addition to cyclophosphamide and dexamethasone. NDMM participants will be randomly assigned (by chance, like flipping a coin) to one of two treatment groups and RRMM participants will be assigned to a third group:

* NDMM - ixazomib (MLN9708) 4.0 mg + cyclophosphamide 300 mg/m^2 + dexamethasone 40 mg
* NDMM - ixazomib (MLN9708) 4.0 mg + cyclophosphamide 400 mg/m^2 + dexamethasone 40 mg
* RRMM - ixazomib (MLN9708) 4.0 mg + cyclophosphamide 300 mg/m^2 + dexamethasone 40 mg

The study enrolled 148 participants. This multi-centre trial will be conducted in the United States, European Union, and Australia.

ELIGIBILITY:
Inclusion Criteria:

Each participant with newly diagnosed multiple myeloma (NDMM) must meet all of the following inclusion criteria to be enrolled in the study:

1. Adult male or female participants 18 years of age or older with a confirmed diagnosis of symptomatic multiple myeloma (MM) according to standard criteria.
2. Participants for whom cyclophosphamide and dexamethasone treatment is appropriate and who are considered not eligible for high-dose therapy (HDT)-stem cell transplantation (SCT) for 1 or more of the following reasons:

   * The participant is 65 years of age or older.
   * The participant is less than 65 years of age but has significant comorbid condition(s) that are, in the opinion of the investigator, likely to have a negative impact on tolerability of HDT-SCT.

Each participant with relapsed and/or refractory multiple myeloma (RRMM) must meet all of the following inclusion criteria to be enrolled in the study:

1. Adult male or female participants 18 years or older with a confirmed diagnosis of symptomatic MM either currently or at the time of initial diagnosis, according to standard criteria, and relapsed and/or refractory disease after 1 to 3 lines of prior therapy. A participant is considered to have refractory disease if disease progression occurred during the treatment period or within 60 days of receiving the last dose of a given therapy. A line of therapy is defined as 1 or more cycles of a single-agent or combination therapy or a sequence of planned treatments such as induction therapy followed by autologous stem cell transplantation (ASCT) and then maintenance therapy.
2. No evidence of graft-versus-host disease for participants who have undergone prior allogeneic stem cell transplantation.

In addition, all participants (NDMM and RRMM) must meet all of the remaining criteria:

1. Participants must have measurable disease defined by at least 1 of the following 3 measurements:

   * Serum M-protein ≥ 1 g/dL (≥ 10 g/L).
   * Urine M-protein ≥ 200 mg/24 hours.
   * Serum free light chain assay: involved free light chain level ≥ 10 mg/dL (≥ 100 mg/L), provided that the serum free light chain ratio is abnormal.
2. Participants must meet all of the following clinical laboratory criteria:

   * Absolute neutrophil count (ANC) ≥ 1000/mm^3 and platelet count ≥ 75,000/mm^3. Platelet transfusions to help participants meet eligibility criteria are not allowed within 3 days prior to administration of the study drug.
   * Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN).
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.
   * Calculated creatinine clearance (CrCL) ≥ 30 mL/min.
3. Eastern Cooperative Oncology Group performance status of 0, 1, or 2.
4. Female participants who:

   * are postmenopausal for at least 1 year before the screening visit, or
   * are surgically sterile, or
   * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 90 days after the last dose of study drug, or
   * agree to practice true abstinence over the period previously described, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [ie, calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.), and
   * adhere to any treatment-specific pregnancy prevention guidelines for cyclophosphamide and dexamethasone.
5. Male participants, even if surgically sterilized (ie, status post-vasectomy), who:

   * agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, or
   * agree to practice true abstinence over the period previously described, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception.), and
   * adhere to any treatment-specific pregnancy prevention guidelines for cyclophosphamide and dexamethasone.
6. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
7. Suitable venous access for the study-required blood sampling.
8. Is willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Prior treatment for multiple myeloma with either standard of care treatment or investigational regimen (for participants with NDMM only).

   NOTE: Prior treatment with corticosteroids (maximum dose of corticosteroids should not exceed the equivalent of 160 mg of dexamethasone over 14 days. Localized radiation is permitted as long as it is below a therapeutic level and administered at least 14 days prior to the first dose of study treatment.
2. Diagnosis of smoldering MM, Waldenström's macroglobulinemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes) syndrome, plasma cell leukemia, primary amyloidosis, myelodysplastic syndrome, or myeloproliferative syndrome.
3. Central nervous system involvement.
4. Diagnosed or treated for another malignancy within 2 years before the first dose or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
5. Peripheral neuropathy Grade 1 with pain or Grade 2 or higher peripheral neuropathy of any cause on clinical examination during the Screening period.
6. Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of study drug, including difficulty swallowing.
7. Infection requiring intravenous (IV) antibiotic therapy or other serious infection within 14 days before the first dose of study drug.
8. Ongoing or active infection, known human immunodeficiency virus (HIV) positive, active hepatitis B or C infection.
9. Systemic treatment with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort within 14 days before the first dose of study treatment.
10. Known allergy to any of the study medications, their analogues, or excipients in the various formulations.
11. Major surgery within 14 days before the first dose of study drug. (Note: kyphoplasty or vertebroplasty is not considered major surgery.)
12. Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the Screening period.
13. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
14. Comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the participant inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
15. Treatment with any investigational products for reasons other than MM within 30 days before the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-03-05 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (24):
- United States (6):
  - Hazard, Kentucky
  - Boston, Massachusetts
  - Rochester, Minnesota
  - St Louis, Missouri
  - New Brunswick, New Jersey
  - Rochester, New York
- Australia (6):
  - Camperdown, New South Wales
  - Concord, New South Wales
  - Waratah, New South Wales
  - Adelaide, South Australia
  - Heidelberg, Victoria
  - Melbourne, Victoria
- Greece (4):
  - Athens, Attica
  - Athens
  - Pátrai
  - Thessaloniki
- Poland (5):
  - Lublin, Lublin Voivodeship
  - Warsaw, Masovian Voivodeship
  - Chorzów
  - Gdansk
  - Lodz
- Sweden (3):
  - Helsingborg, Skåne County
  - Stockholm, Södermanland County
  - Lund

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Dimopoulos MA, Grosicki S, Jedrzejczak WW, Nahi H, Gruber A, Hansson M, Gupta N, Byrne C, Labotka R, Teng Z, Yang H, Grzasko N, Kumar S. All-oral ixazomib, cyclophosphamide, and dexamethasone for transplant-ineligible patients with newly diagnosed multiple myeloma. Eur J Cancer. 2019 Jan;106:89-98. doi: 10.1016/j.ejca.2018.09.011. Epub 2018 Nov 22. PMID 30471652
- [Derived] Kumar SK, Grzasko N, Delimpasi S, Jedrzejczak WW, Grosicki S, Kyrtsonis MC, Spencer A, Gupta N, Teng Z, Byrne C, Labotka R, Dimopoulos MA. Phase 2 study of all-oral ixazomib, cyclophosphamide and low-dose dexamethasone for relapsed/refractory multiple myeloma. Br J Haematol. 2019 Feb;184(4):536-546. doi: 10.1111/bjh.15679. Epub 2018 Nov 20. PMID 30460684

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 23 investigative sites in Australia, Greece, Poland, Sweden and the United States from 05 March 2014 to 29 June 2018.
Pre-assignment Details: Participants with NDMM were enrolled in 1 of 2 arms to receive 4.0 mg ixazomib in combination with 300 or 400 mg cyclophosphamide and 40 mg dexamethasone (CCd); participants with RRMM were enrolled in 1 arm to receive ixazomib 4.0 mg CCd. All arms included a safety lead-in cohort for pharmacokinetics (PK) analysis.
Groups:
- Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM): Ixazomib 4.0 mg, capsules, orally, on Days 1, 8, 15 of a 28-day cycle and cyclophosphamide (CYC) 300 mg/m^2, tablets, orally, on Days 1, 8 and 15 of a 28-day cycle and dexamethasone (DEX) 40 mg, tablets, orally, on Days 1, 8, 15 and 22 (dose reduced to 20 mg for patients >75 years) of a 28-day cycle until PD/death or unacceptable toxicity in participants with RRMM.
Period: Overall Study
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM)
Started | 36 | 34 | 78
Completed (Completed=Completed Study Treatment) | 4 | 6 | 8
Not Completed | 32 | 28 | 70
Not completed — Progressive Disease | 18 | 11 | 40
Not completed — Adverse Event | 8 | 10 | 17
Not completed — Withdrawal by Subject | 1 | 2 | 6
Not completed — Study Terminated by Sponsor | 1 | 1 | 1
Not completed — Reason not Specified | 4 | 4 | 6

BASELINE CHARACTERISTICS:
Population: Safety population was defined as all participants who received at least 1 dose of any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM) | Total
Number analyzed (Participants) | 36 | 34 | 78 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.4 (5.48) | 74.1 (5.80) | 63.5 (9.85) | 68.3 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37 | 74
  Male | 15 | 18 | 41 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 35 | 33 | 75 | 143
  Unknown or Not Reported | 0 | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 35 | 34 | 74 | 143
  Other | 1 | 0 | 2 | 3
  Asian | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 1 | 1
Height [Mean (Standard Deviation); unit: centimeters (cm)] — Population: Number Analyzed is the number of participants with data available for analysis.
  centimeters (cm)
    number analyzed (Participants) | 36 | 34 | 77 | 147
    (all) | 163.5 (11.35) | 163.5 (12.47) | 165.9 (10.47) | 164.8 (11.16)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 73.6 (11.8) | 73.0 (17.54) | 78.1 (16.80) | 75.8 (15.99)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: meters squared (m^2)] — BSA = square root (height(cm) x weight (kg) / 3600.
  meters squared (m^2) | 1.8 (0.17) | 1.8 (0.26) | 1.9 (0.23) | 1.8 (0.23)

OUTCOME MEASURES:

1. Primary Outcome: Combined Response Rate During the Induction Phase in Newly Diagnosed Multiple Myeloma (NDMM) Participants
Description: Combined Response Rate is the percentage of participants with Complete Response (CR), including stringent Complete Response (sCR), and Very Good Partial Response (VGPR) according to the International Myeloma Working Group (IMWG) criteria during the Induction Phase (Cycles 1-13, 28-day cycles). CR=negative immunofixation of serum and urine, disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow. VGPR=serum and urine M-component detectable by immunofixation but not on electrophoresis or 90% reduction in serum M-component plus urine M-component <100 mg/24 hour.
Time Frame: Day 1 of Cycles 1-13, 28-day cycles (Up to 1 year)
Population: Response Evaluable Population was defined as participants who received at least 2 of the 3 ixazomib doses during Cycle 1, had measurable disease at Baseline, and at least 1 postbaseline response assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM)
Number analyzed (Participants) | 33 | 34
percentage of participants | 27 [13 to 46] | 24 [11 to 41]
Statistical Analysis 1: Comparison: Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM); P-value tests the null hypothesis: CR+VGPR rate=27% in treatment arms obtained using the one-sided Chi-Square test with alpha=0.10; Test type: Other; p = 0.4859, Chi-squared
Statistical Analysis 2: Comparison: Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.6757, Chi-squared

2. Primary Outcome: Overall Response Rate (ORR) in Relapsed and/or Refractory Multiple Myeloma (RRMM) Participants
Description: ORR is the percentage of participants with CR, VGPR or PR according to IMWG criteria. CR=negative immunofixation of serum and urine, disappearance of any soft tissue plasmacytomas and <5% plasma cells (PC) in bone marrow. VGPR=serum and urine M-component detectable by immunofixation but not on electrophoresis or 90% reduction in serum M-component plus urine M-component <100 mg/24 hour. PR=50% reduction of serum M-protein and reduction in 24 hour urine M-protein by 90% or <200 mg/24 hour or decrease 50% difference between involved free light chain (FLC) levels or 50% reduction in bone marrow plasma cells if baseline percentage was 30%; and if present at Baseline, 50% reduction in the size of soft tissue plasmacytomas.
Time Frame: Day 1 of each 28 day cycle (Up to 45 months)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM)
Number analyzed (Participants) | 73
percentage of participants | 49 [37 to 61]
Statistical Analysis 1: Comparison: Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM); P-value tests the null hypothesis: CR+VGPR+PR rate=60% obtained using the one-sided Chi-Square test with alpha=0.10; Test type: Other; p = 0.9688, Chi-squared

3. Secondary Outcome: Number of Participants With Adverse Events (AEs), Grade 3 or Higher AEs, AEs Resulting in Treatment Discontinuation, AEs Resulting in Dose Reduction and Serious Adverse Events (SAEs) in NDMM Participants
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. This includes any newly occurring event, or a previous condition that has increased in severity or frequency since the administration of study drug.
  A SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is a medically important event. Relationship of each AE to study drug was determined by the Investigator.
Time Frame: First dose of study drug through 30 days after last dose of drug (Up to 45 months)
Population: Safety Population was defined as all participants who receive at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM)
Number analyzed (Participants) | 36 | 34
Participants
  Any AE | 35 | 34
  Grade 3 or Higher AEs | 27 | 27
  AEs Resulting in Treatment Discontinuation | 9 | 11
  AEs Resulting in Dose Reduction | 11 | 10
  SAEs | 17 | 20

4. Secondary Outcome: Percentage of Participants With CR + VGPR + PR (ORR), CR, VGPR, PR and Stable Disease (SD), Progressive Disease (PD) During the Induction Phase
Description: Percentage of participants with CR + VGPR + PR (ORR), CR, VGPR, PR, SD, PD according to IMWG criteria. CR=negative immunofixation of serum and urine; disappearance of soft tissue plasmacytomas;<5% PC in bone marrow. VGPR=serum and urine M-component detectable by immunofixation but not on electrophoresis or 90% reduction in serum M-component plus urine M-component <100 mg/24 hour. PR=50% reduction of serum M-protein and reduction in 24 hour urine M-protein by 90% or <200 mg/24 hour or decrease 50% difference between involved FLC levels or 50% reduction in bone marrow plasma cells if baseline percentage was 30%; and if present at Baseline, 50% reduction in the size of soft tissue plasmacytomas. SD=not meeting criteria for VGPR, PR or PD. PD=25% increase in lowest value any of the following: serum M-component, urine M-component, difference between involved and uninvolved FLC levels, bone marrow PC percentage; new or increase in size of existing bone lesions or soft tissue plasmacytomas.
Time Frame: Day 1 of Cycles 1-13, 28-day cycles (Up to 1 year)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM)
Number analyzed (Participants) | 33 | 34
percentage of participants
  CR + VGPR + PR | 79 [61 to 91] | 71 [53 to 85]
  CR | 12 [3 to 28] | 9 [2 to 24]
  VGPR | 15 [5 to 32] | 15 [5 to 31]
  PR | 67 [48 to 82] | 62 [44 to 78]
  SD | 12 [3 to 28] | 18 [7 to 35]
  PD | 0 [0 to 0] | 3 [1 to 15]

5. Secondary Outcome: Percentage of Participants With CR + VGPR + PR (ORR), CR + VGPR, CR, VGPR, PR, SD and PD Throughout the Entire Treatment Period in NDMM Participants
Description: as for outcome 4
Time Frame: Day 1 of each 28-day Cycle (Up to 45 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM)
Number analyzed (Participants) | 33 | 34
percentage of participants
  CR + VGPR + PR | 82 [65 to 93] | 71 [53 to 85]
  CR + VGPR | 36 [20 to 55] | 32 [17 to 51]
  CR | 15 [5 to 32] | 12 [3 to 27]
  VGPR | 21 [9 to 39] | 21 [9 to 38]
  PR | 67 [48 to 82] | 59 [41 to 75]
  SD | 18 [7 to 35] | 18 [7 to 35]
  PD | 0 [0 to 0] | 6 [1 to 20]

6. Secondary Outcome: Time to Response (TTR) in NDMM Participants During the Induction Phase
Description: TTR is defined as the time interval from the date of the first dose of study treatment to the date of the first documented confirmed response of PR or better up to the initiation of alternative therapy in a participant who responded.
Time Frame: Up to 1 year
Population: Participants from the Response Evaluable Population, defined as participants who received at least 2 of the 3 ixazomib doses during Cycle 1, had measurable disease at Baseline, and at least 1 postbaseline response assessment, who responded.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM)
Number analyzed (Participants) | 26 | 23
months | 2.2 [0.95 to 2.92] | 1.9 [0.95 to 1.9]

7. Secondary Outcome: Duration of Response (DOR) in NDMM Participants
Description: DOR is defined as the time from the date of first documentation of a confirmed PR or better to the date of first documented PD up to the initiation of alternative therapy.
Time Frame: Up to 45 Months
Population: Participants from the Response Evaluable Population, participants who received at least 2 of the 3 ixazomib doses during Cycle 1, had measurable disease at Baseline and at least 1 postbaseline response assessment, who responded. Responders without PD were censored at the date of SD or better prior to the date of alternative therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM)
Number analyzed (Participants) | 26 | 23
months | 32.2 [18.66 to NA] — 95% Confidence Interval (CI) Upper Limit was not estimable due to the low number of participants with events. | 36.6 [19.75 to NA] — 95% CI Upper Limit was not estimable due to the low number of participants with events.

8. Secondary Outcome: Time to Progression (TTP) in NDMM Participants
Description: TTP is defined as the time from the date of first dose of study treatment to the date of first documentation of disease progression.
Time Frame: Up to 45 months
Population: Safety Population was defined as all participants who received at least 1 dose of any study drug. Participants without documentation of PD were censored at the date of last response assessment that is SD or better prior to the date of the alternative therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM)
Number analyzed (Participants) | 36 | 34
months | 30.9 [19.58 to 41.66] | 32.2 [20.27 to NA] — 95% CI Upper Limit was not estimable due to the low number of participants with events.

9. Secondary Outcome: Progression Free Survival (PFS) in NDMM Participants
Description: PFS is defined as the time from the date of first dose of study treatment to the date of the first documented disease progression or death.
Time Frame: Up to 45 months
Population: Safety Population was defined as all participants who received at least 1 dose of any study drug. Participants without documentation of PD or death were censored at the date of last response assessment that is SD or better prior to the date of the alternative therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM)
Number analyzed (Participants) | 36 | 34
months | 23.5 [15.67 to 39.59] | 23.0 [15.90 to NA] — 95% CI Upper Limit was not estimable due to the low number of participants with events.

10. Secondary Outcome: Number of Participants With AEs, SAEs, AEs Resulting in Discontinuation and AEs Resulting in Dose Reduction in NDMM Participants Remaining on Treatment After 13 Cycles
Description: as for outcome 3
Time Frame: First dose of study drug through 30 days after the last dose of drug (Up to 45 months)
Population: Safety Population was defined as all participants who receive at least 1 dose of any study drug. Number of participants analyzed is the number of participants who remained on treatment after 13 cycles.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM)
Number analyzed (Participants) | 24 | 22
Participants
  Any AE | 22 | 20
  SAE | 6 | 4
  AEs Resulting in Treatment Discontinuation | 1 | 2
  AEs Resulting in Dose Reduction | 5 | 4

11. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) During the Induction Phase in NDMM Participants
Description: EORTC QLQ-C30 is a patient completed 30 item questionnaire that consists of 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The patient evaluates their health status over the previous week. There are 28 questions answered on a 4-point scale where1=Not at all (best) to 4=Very Much (worst) and 2 questions answered on a 7-point scale where 1=Very poor (worst) to 7= Excellent (best). All of the scales and single-item measures are transformed to a score:0 to 100. For functioning scales and global QOL higher scores indicate better functioning (a positive change from Baseline indicates improvement); for symptom scales higher scores indicate more severe symptoms (a negative change from Baseline indicates improvement).
Time Frame: Baseline (BL) (Day 1 of Cycle 1), Day 1 of Cycle 13 (Up to 1 year)
Population: Participants from the Safety Population, defined as all participants who received at least 1 dose of any study drug, with data available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM)
Number analyzed (Participants) | 24 | 23
score on a scale
  Global Health Status/QoL, Change from BL; Cycle 13 | 3.47 (30.783) | -5.43 (24.180)
  Physical functioning, Change from BL at Cycle 13 | 14.17 (35.675) | 17.97 (20.640)
  Role functioning, Change from BL at Cycle 13 | 8.33 (43.127) | 6.52 (35.441)
  Emotional functioning, Change from BL at Cycle 13 | 11.34 (27.837) | 2.54 (15.977)
  Cognitive functioning, Change from BL at Cycle 13 | 2.78 (22.877) | -7.25 (14.058)
  Social functioning, Change from BL at Cycle 13 | 9.03 (39.921) | -11.59 (29.914)
  Fatigue, Change from BL at Cycle 13 | -10.88 (35.307) | -6.76 (30.473)
  Nausea/Vomiting, Change from BL at Cycle 13 | -4.86 (26.228) | -4.35 (19.603)
  Pain, Change from BL at Cycle 13 | -13.89 (52.628) | -10.87 (39.443)
  Dyspnea, Change from BL at Cycle 13 | -11.11 (37.644) | -7.25 (40.147)
  Insomnia, Change from BL at Cycle 13 | -16.67 (46.104) | -10.14 (35.441)
  Appetite Loss, Change from BL at Cycle 13 | -18.06 (42.822) | -7.25 (24.529)
  Constipation, Change from BL at Cycle 13 | -13.89 (39.215) | -5.80 (41.013)
  Diarrhea, Change from BL at Cycle 13 | -2.78 (30.954) | 5.80 (19.207)
  Financial Difficulties, Change from BL at Cycle 13 | 4.17 (26.580) | 1.45 (30.942)

12. Secondary Outcome: Percentage of Participants With CR + VGR + PR (ORR), CR, VGPR, and PR in NDMM Participants Remaining on Treatment After 13 Cycles
Description: Percentage of participants with Overall Response (CR + VGPR + PR), CR, VGPR and PR according to IMWG criteria. CR=negative immunofixation of serum and urine; disappearance of soft tissue plasmacytomas;<5% PC in bone marrow. VGPR=serum and urine M-component detectable by immunofixation but not on electrophoresis or 90% reduction in serum M-component plus urine M-component <100 mg/24 hour. PR=50% reduction of serum M-protein and reduction in 24 hour urine M-protein by 90% or <200 mg/24 hour or decrease 50% difference between involved FLC levels or 50% reduction in bone marrow plasma cells if baseline percentage was 30%; and if present at Baseline, 50% reduction in the size of soft tissue plasmacytomas.
Time Frame: Day 1 of each 28-day Cycle (Up to 45 months)
Population: Participants from the Response Evaluable Population, participants who received at least 2 of the 3 ixazomib doses during Cycle 1, had measurable disease at Baseline and at least 1 postbaseline response assessment, with both an Induction and Maintenance response.
Measure: Number; unit: percentage of participants
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM)
Number analyzed (Participants) | 24 | 21
percentage of participants
  CR + VGPR + PR | 75.0 | 85.7
  CR | 16.7 | 19.0
  VGPR | 20.8 | 28.6
  PR | 37.5 | 38.1

13. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Ixazomib in NDMM Participants
Time Frame: Cycle 1 Days 1 and 15 predose and at multiple timepoints (up to 168 hours) postdose
Population: PK-Evaluable Population was defined as participants in the safety lead-in cohort who have sufficient dosing data and ixazomib concentration-time data to permit calculation of PK parameters. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: nanogram/mL (ng/mL)
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM)
Number analyzed (Participants) | 6 | 6
nanogram/mL (ng/mL)
  Cycle 1 Day 1 | 64.283 (36.283) | 46.600 (34.7722)
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 5
  Cycle 1 Day 15 | 53.145 (46.3782) | 62.280 (39.4249)

14. Secondary Outcome: Tmax: Time to First Occurrence of Cmax for Ixazomib in NDMM Participants
Time Frame: Cycle 1 Days 1 and 15 predose and at multiple timepoints (up to 168 hours) postdose
Population: as for outcome 13
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM)
Number analyzed (Participants) | 6 | 6
hour (hr)
  Cycle 1 Day 1 | 1.250 [0.92 to 1.58] | 1.040 [0.50 to 2.00]
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 5
  Cycle 1 Day 15 | 1.000 [0.45 to 4.00] | 1.000 [0.50 to 1.50]

15. Secondary Outcome: AUCtau: Area Under the Concentration-time Curve During a Dosing Interval for Ixazomib in NDMM Participants
Time Frame: Cycle 1 Days 1 and 15 predose and at multiple timepoints (up to 168 hours) postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM)
Number analyzed (Participants) | 6 | 6
hr*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 5
  Cycle 1 Day 1 | 885.167 (354.1465) | 792.600 (650.5665)
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 5
  Cycle 1 Day 15 | 1338.333 (746.2902) | 1226.600 (527.5792)

16. Secondary Outcome: Number of Participants With AEs, Grade 3 or Higher AEs, AEs Resulting in Treatment Discontinuation, AEs Resulting in Dose Reduction, SAEs in RRMM Participants
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment.
  A SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is a medically important event. Relationship of each AE to study drug was determined by the Investigator.
Time Frame: First dose of study drug through 30 days after last dose of drug (Up to 45 months)
Population: Safety population was defined as all participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM)
Number analyzed (Participants) | 78
Participants
  Any AE | 72
  Grade 3 or Higher AE | 49
  AEs Resulting in Treatment Discontinuation | 19
  AEs Resulting in Dose Reduction | 30
  SAEs | 30

17. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Ixazomib in RRMM Participants
Time Frame: Cycle 1 Days 1 and 15 predose and at multiple timepoints (up to 168 hours) postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM)
Number analyzed (Participants) | 7
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 6
  Cycle 1 Day 1 | 47.400 (36.7083)
  Cycle 1 Day 15 | 52.229 (39.6006)

18. Secondary Outcome: Tmax: Time to First Occurrence of Cmax for Ixazomib in RRMM Participants
Time Frame: Cycle 1 Days 1 and 15 predose and at multiple timepoints (up to 168) hours postdose
Population: as for outcome 13
Measure: Median (Full Range); unit: hr
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM)
Number analyzed (Participants) | 7
hr
  Cycle 1 Day 1: number analyzed (Participants) | 6
  Cycle 1 Day 1 | 1.225 [0.50 to 3.42]
  Cycle 1 Day 15 | 2.000 [0.50 to 8.00]

19. Secondary Outcome: AUCtau: Area Under the Concentration-time Curve During a Dosing Interval for Ixazomib in RRMM Participants
Time Frame: Cycle 1 Days 1 and 15 predose and at multiple timepoints (up to 168 hours) postdose
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM)
Number analyzed (Participants) | 7
hr*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 6
  Cycle 1 Day 1 | 518.167 (78.8274)
  Cycle 1 Day 15 | 1241.000 (657.4978)

20. Secondary Outcome: Percentage of Participants With (CR + VGPR), CR, VGPR, PR, SD and PD in RRMM Participants
Description: as for outcome 4
Time Frame: Day 1 of each 28-day Cycle (Up to 45 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM)
Number analyzed (Participants) | 73
percentage of participants
  CR + VGPR | 19 [11 to 30]
  CR | 5 [2 to 13]
  VGPR | 14 [7 to 24]
  PR | 44 [32 to 56]
  SD | 37 [26 to 49]
  PD | 10 [4 to 19]

21. Secondary Outcome: Time to Response (TTR) in RRMM Participants
Description: TTR is defined as the time interval from the date of the first dose of study treatment to the date of the first documented confirmed response of PR or better up to the alternative therapy in a participant who responded.
Time Frame: Up to 45 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM)
Number analyzed (Participants) | 36
months | 2.1 [0.95 to 3.12]

22. Secondary Outcome: Duration of Response (DOR) in RRMM Participants
Description: DOR is defined as the time from the date of first documentation of a confirmed PR or better to the date of first documented PD up to the alternative therapy.
Time Frame: Up to 45 months
Population: Participants from the Response Evaluable Population, participants who received at least 2 of the 3 ixazomib doses during Cycle 1, had measurable disease at Baseline and at least 1 postbaseline response assessment, who responded. Responders without PD were censored at the date of SD or better prior to the date of the alternative therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM)
Number analyzed (Participants) | 36
months | 26.3 [12.22 to NA] — 95% CI Upper Limit was not estimable due to the low number of participants with events.

23. Secondary Outcome: Time to Progression (TTP) in RRMM Participants
Description: as for outcome 8
Time Frame: Up to 45 months
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM)
Number analyzed (Participants) | 78
months | 16.8 [11.30 to 24.67]

24. Secondary Outcome: Progression Free Survival (PFS) in RRMM Participants
Description: as for outcome 9
Time Frame: Up to 45 months
Population: Safety Population was defined as all participants who received at least 1 dose of any study drug. Participants without documentation of PD or death were censored at the date of last response assessment that was SD or better prior to the date of the alternative therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM)
Number analyzed (Participants) | 78
months | 14.2 [9.69 to 20.57]

25. Secondary Outcome: Change From Baseline in EORTC Quality of Life Questionnaire (QLQ-C30) in RRMM Participants
Description: as for outcome 11
Time Frame: Baseline (Day 1 of Cycle 1), Day 1 of End of Treatment (EOT) (Up to 45 months)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM)
Number analyzed (Participants) | 50
score on a scale
  Global Health Status/QoL, Change from BL at EOT | -5.50 (20.798)
  Physical functioning, Change from BL at EOT | -6.00 (19.806)
  Role functioning, Change from BL at EOT | -7.67 (30.344)
  Emotional functioning, Change from BL at EOT | -5.00 (23.023)
  Cognitive functioning, Change from BL at EOT | -5.33 (19.760)
  Social functioning, Change from BL at EOT | -11.33 (26.177)
  Fatigue, Change from BL at EOT | 5.11 (22.695)
  Nausea/Vomiting, Change from BL at EOT | 3.33 (14.677)
  Pain, Change from BL at EOT | 5.00 (28.621)
  Dyspnea, Change from BL at EOT | 10.00 (27.970)
  Insomnia, Change from BL at EOT | -6.00 (27.512)
  Appetite Loss, Change from BL at EOT | 4.67 (24.290)
  Constipation, Change from BL at EOT | 2.00 (18.332)
  Diarrhea, Change from BL at EOT | 6.00 (19.852)
  Financial Difficulties, Change from BL at EOT | 4.00 (20.909)

ADVERSE EVENTS:
Time Frame: First dose of study drug through 30 days after last dose of drug (Up to 45 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM) | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM)
All-Cause Mortality (participants affected / at risk) | 3/36 | 2/34 | 5/78
Serious Adverse Events (participants affected / at risk) | 17/36 | 20/34 | 30/78
Other Adverse Events (participants affected / at risk) | 34/36 | 34/34 | 69/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) (N=36) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM) (N=34) | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM) (N=78)
Pneumonia (Infections and infestations) | 4 | 2 | 3 — One treatment-emergent death occurred during treatment with Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM) and is not related.
Bronchitis (Infections and infestations) | 0 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM) and is related.
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) and is not related.
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Rectal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 — One treatment-emergent (TE) death occurred during treatment with Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM) and is not related.
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 — 1 TE death occurred during treatment with Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM), 1 with Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM) and 1 with Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM) and all 3 are not related.
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) and is not related.
Pyrexia (General disorders) | 1 | 1 | 2
Fatigue (General disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM) and is related.
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM) and is not related.
Syncope (Nervous system disorders) | 1 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Pemphigus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Light chain analysis increased (Investigations) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (NDMM) (N=36) | Ixazomib 4.0 mg + CYC 400 mg/m^2 + DEX 40 mg (NDMM) (N=34) | Ixazomib 4.0 mg + CYC 300 mg/m^2 + DEX 40 mg (RRMM) (N=78)
Upper respiratory tract infection (Infections and infestations) | 9 | 3 | 21
Bronchitis (Infections and infestations) | 5 | 4 | 12
Nasopharyngitis (Infections and infestations) | 5 | 4 | 6
Respiratory tract infection (Infections and infestations) | 3 | 4 | 8
Herpes zoster (Infections and infestations) | 6 | 3 | 5
Influenza (Infections and infestations) | 3 | 0 | 6
Conjunctivitis (Infections and infestations) | 2 | 1 | 5
Urinary tract infection (Infections and infestations) | 2 | 3 | 3
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 5
Pharyngitis (Infections and infestations) | 2 | 1 | 3
Pneumonia (Infections and infestations) | 1 | 1 | 4
Oral herpes (Infections and infestations) | 2 | 0 | 3
Cellulitis (Infections and infestations) | 2 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 11 | 9 | 26
Nausea (Gastrointestinal disorders) | 8 | 10 | 19
Vomiting (Gastrointestinal disorders) | 6 | 9 | 9
Constipation (Gastrointestinal disorders) | 8 | 7 | 8
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 6
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 4
Flatulence (Gastrointestinal disorders) | 0 | 0 | 4
Gastritis (Gastrointestinal disorders) | 2 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 11 | 11 | 19
Neutropenia (Blood and lymphatic system disorders) | 6 | 16 | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 4 | 18
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 4
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1
Fatigue (General disorders) | 8 | 7 | 15
Oedema peripheral (General disorders) | 8 | 9 | 5
Pyrexia (General disorders) | 4 | 6 | 4
Influenza like illness (General disorders) | 1 | 1 | 4
Non-cardiac chest pain (General disorders) | 1 | 1 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 10 | 10
Dizziness (Nervous system disorders) | 3 | 2 | 7
Hypoaesthesia (Nervous system disorders) | 4 | 3 | 5
Headache (Nervous system disorders) | 3 | 3 | 3
Neuropathy peripheral (Nervous system disorders) | 4 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 6 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 2 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 6
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 3 | 10
Anxiety (Psychiatric disorders) | 1 | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 2 | 1
Hypertension (Vascular disorders) | 2 | 7 | 2
Hypotension (Vascular disorders) | 1 | 2 | 2
Weight decreased (Investigations) | 4 | 3 | 1
Blood creatinine increased (Investigations) | 3 | 2 | 0
Cataract (Eye disorders) | 0 | 2 | 5
Glaucoma (Eye disorders) | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 3 | 3
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT02046070/SAP_000.pdf
  • Study Protocol (2014-05-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT02046070/Prot_001.pdf